CLINICAL TRIAL: NCT01878916
Title: Plasma Cobalamin, Folate, Pyridoxine and Homocysteine Levels and Thrombosis in Patients With Philadelphia-chromosome-negative Myeloproliferative Neoplasms
Brief Title: Plasma Vitamin and Homocysteine Levels and Thrombosis in Patients With Ph-negative MPNs
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. A. Emre Eşkazan, MD, Istanbul University
Other Study IDs: HcyMPN
Record Dates: First submitted 2013-05-29; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Thrombosis
Keywords: the incidence of thrombosis,; the effect of Hcy on thrombosis formation,; the relation between Hcy and plasma vitamin levels,; to compare these results with the control group
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Hyperhomocysteinemia is a risk for thrombosis. Thrombosis is more frequent in myeloproliferative neoplasms (MPNs) than the normal population. In this study, we investigated the thrombosis incidence, the effects of plasma homocysteine levels on thrombosis, and the correlations between folate, cobalamin, pyridoxine and homocysteine levels in MPNs, and to compare these results with the healthy controls.

DETAILED DESCRIPTION:
Thirty-one new or formerly diagnosed MPN patients who consecutively visitted our outpatient clinic, as well as 40 age and sex matched healthy controls were enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

Adult MPN patients and healthy controls who gave a written consent were included in the study.

Exclusion Criteria:

Exclusion criteria included not giving a written consent and using medications without an indication which may have an effect on plasma homocysteine and vitamin levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between January and June 2003, thirty-one new or formerly diagnosed MPN patients who consecutively visitted our clinic, as well as 40 age and sex matched healthy controls were enrolled in this study.
Sampling Method: Probability Sample
Dates: Start 2003-01; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Thrombosis | at least 1 year

SECONDARY OUTCOMES:
High Hcy level | 1 year

OTHER OUTCOMES:
Death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Emre Eskazan, MD, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)